CLINICAL TRIAL: NCT00577317
Title: A Prospective Randomized Single Blind Phase III Trial Comparing Flexitouch Home Maintenance Therapy to Standard Home Maintenance Therapy for Lower Extremity Lymphedema Resulting From Treatment of Gynecologic Malignancy
Brief Title: Flexitouch® Home Maintenance Therapy or Standard Home Maintenance Therapy in Treating Patients With Lower-Extremity Lymphedema Caused by Treatment for Cervical Cancer, Vulvar Cancer, or Endometrial Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GOG-0236; NCI-2009-00602 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000579834; GOG-0236 (Other: Gynecologic Oncology Group); GOG-0236 (Other: DCP); GOG-0236 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Lymphedema; Stage 0 Cervical Cancer; Stage 0 Uterine Corpus Cancer; Stage 0 Vulvar Cancer; Stage I Uterine Corpus Cancer; Stage I Vulvar Cancer; Stage IA Cervical Cancer; Stage IB Cervical Cancer; Stage II Uterine Corpus Cancer; Stage II Vulvar Cancer; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage III Uterine Corpus Cancer; Stage III Vulvar Cancer; Stage IV Uterine Corpus Cancer; Stage IVA Cervical Cancer; Stage IVB Cervical Cancer; Stage IVB Vulvar Cancer
MeSH Terms: conditions — Lymphedema; Uterine Cervical Dysplasia; Vulvar Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Arm 1 (Experimental): Patients receive standard home maintenance therapy and perform self-manual lymphatic drainage once daily for 60 minutes for 24 weeks.
  Interventions: Procedure: Management of Therapy Complications; Other: Quality-of-Life Assessment
- Arm II (Experimental): Patients receive Flexitouch® home maintenance therapy once daily for 60 minutes for 24 weeks
  Interventions: Procedure: Management of Therapy Complications; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Management of Therapy Complications — Receive standard home maintenance therapy and perform self-manual lymphatic drainage
  Other Names: complications of therapy, management of
  Arms: Arm 1
Procedure: Management of Therapy Complications — Receive Flexitouch home maintenance therapy
  Other Names: complications of therapy, management of
  Arms: Arm II
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial is studying Flexitouch® home maintenance therapy to see how well it works compared with standard home maintenance therapy in treating patients with lower-extremity lymphedema caused by treatment for cervical cancer, vulvar cancer, or endometrial cancer. Flexitouch® home maintenance therapy may lessen lower-extremity lymphedema caused by treatment for gynecologic cancer. It is not yet known whether the Flexitouch® system is more effective than standard home maintenance therapy in treating lymphedema.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare the effectiveness of the Flexitouch® System to standard home lymphedema therapy (Manual Lymphatic Drainage) in the management of lower-extremity lymphedema in women with a history of cervical, vulvar, or endometrial cancer.

SECONDARY OBJECTIVE:

I. Compare the quality of life (QOL) and functional status between patients using the Flexitouch® System and those following standard home lymphedema treatment (Manual Lymphatic Drainage) programs in the management of lower-extremity lymphedema

OUTLINE: This is a multicenter study. Patients are stratified according to site of cancer (cervical vs vulvar vs endometrial) and stage of lymphedema at diagnosis. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive standard home maintenance therapy and perform self-manual lymphatic drainage once daily for 60 minutes for 24 weeks.

ARM II: Patients receive Flexitouch® home maintenance therapy once daily for 60 minutes for 24 weeks.

Clinical staff measure patients' lower limb (both) volumes and patients complete quality of life questionnaires at baseline, every 8 weeks during treatment, and at completion of study treatment.

ELIGIBILITY:
Criteria:

* Has lower-extremity lymphedema on one side of the body caused by surgery, chemotherapy, and/or radiation therapy.
* At least 6 months since clinic therapy for lower-extremity lymphedema
* Is within 3 years from finishing cancer treatment
* No active or recurrent cancer
* More than 3 months since cancer treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-12; Primary Completion 2009-07-27 (Actual); Study Completion 2009-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Levi Downs, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Opened to accrual 12/26/2007 was terminated to enrollment on 7/21/2009 due to poor accrual. Target accrual was 262 patients.
Period: Overall Study
Arm/Group | Arm 1 | Arm II
Started | 0 | 2
Completed | 0 | 0
Not Completed | 0 | 2
Not completed — Study Terminated | 0 | 2

BASELINE CHARACTERISTICS:
Population: Eligible and Evaluable subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm II | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 0 | 0 | 0
  30-39 years | 0 | 1 | 1
  40-49 years | 0 | 0 | 0
  50-59 years | 0 | 0 | 0
  60-69 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Lower-extremity Volumes for Both Unaffected and Affected Legs
Description: Volume for both lower extremities were going to be measured to determine if using the Flexi-touch was a more effective method to control lymphedema. Given that the study closed due to poor accrual (2 participants) analysis was not done.
Time Frame: From registration to study discontinuation. A maximum of 7 months.
Population: Eligible and evaluable participants. There were no evaluable participants due to low accrual.
Arm/Group | Arm 1 | Arm II
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Quality of Life (QOL) and Functional Status as Assessed by the Lymphedema Questionnaire
Description: Quality of life was to be assessed to compare QOL between arms. Due to poor accrual (2 participants) and study closure, data was not collected and analysis was not done. There are no results to report due to the limited number of participants.
Time Frame: From registration to study discontinuation. A maximum of 7 months.
Reporting Status: Not Posted

3. Secondary Outcome: Compliance With Treatment as Assessed by the Number of Days Per Week Using MLD or Flexitouch System and Duration/Day of MLD and Flexitouch System Treatment
Description: Compliance with treatment was to be measured between both arms of the study. Due to poor accrual (2 participants) and study closure, data was not collected and analysis was not done. There are no results to report due to the limited number of participants.
Time Frame: From registration to study discontinuation. A maximum of 7 months.
Reporting Status: Not Posted

4. Secondary Outcome: Pain in Affected Limb
Description: Pain in affected limb was to be measured. Due to poor accrual (2 participants) and study closure, data was not collected and analysis was not done. There are no results to report due to the limited number of participants.
Time Frame: From registration to study discontinuation. A maximum of 7 months.
Reporting Status: Not Posted

5. Secondary Outcome: Incidence of Deep-vein Thrombosis
Description: Incidence of deep-vein thrombosis was to be measured during the study. Unfortunately, due to low accrual study was closed. Analysis will not be performed.
Time Frame: From registration to study discontinuation. A maximum of 7 months.
Reporting Status: Not Posted

6. Secondary Outcome: Incidence of Cellulitis
Description: Incidence of cellulitis in both arms was planned to measured. Due to poor accrual (2 participants) and study closure, data was not collected and analysis was not done. There are no results to report due to the limited number of participants.
Time Frame: From registration to study discontinuation. A maximum of 7 months.
Reporting Status: Not Posted

7. Secondary Outcome: Need for Unscheduled Visits at the Patients' Lymphedema Clinic
Description: The need for unscheduled visits at the patient's lymphedema clinic was going to be analyzed. Due to poor accrual (2 participants) and study closure, data was not collected and analysis was not done. There are no results to report due to the limited number of participants.
Time Frame: From registration to study discontinuation. A maximum of 7 months.
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Two participants enrolled in this study. The study was closed early due to poor accrual.
Arm/Group | Arm 1 | Arm II
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less